CLINICAL TRIAL: NCT05298917
Title: Influence of Silicone Hydrogel Extended Contact Lens Wear on Corneal Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Nosch (Other)
Responsible Party: Sponsor-Investigator, Daniela Nosch, Clinical Professor, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-D0011
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cornea
Keywords: silicone hydrogel contact lens; extended contact lens wear; corneal sensitivity; esthesiometry
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- extended contact lens wear (Other): subjects wear silicone hydrogel contact lenses continuously for 7+/- 1 days - corneal sensitivity will be measured and compared at baseline versus after extended contact lens wear
  Interventions: Device: silicone hydrogel contact lens

INTERVENTIONS:
Device: silicone hydrogel contact lens — silicone hydrogel contact lens

SUMMARY:
Soft contact lens wear reduces the amount of oxygen reaching the eye, which may have an influence on corneal sensitivity. The aim of this study is to measure corneal sensitivity with means of liquid jet esthesiometry at baseline and after 6 days of continuous, extended contact lens wear.

DETAILED DESCRIPTION:
Contact lens wear may have an influence on corneal sensitivity, by three mechanisms: hypoxic, mechanical and inflammatory. Extended silicone hydrogel contact lens wear increases the risk of infections. A change in corneal sensitivity may be considered as an indicator for change in corneal physiology. It is there the aim of this study is to measure corneal sensitivity with means of liquid jet esthesiometry at baseline and after 6 days of continuous, extended contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

* no contact lens wear three days before first visit
* corneal radius between 7.4 and 8.0; if corneal radius >8.0, corneal diameter must be at least 12 mm; if corneal radius < 7.4, corneal diameter must be < 12.0
* OSDI score no higher than 13 points

Exclusion Criteria:

* systemic disease that may have an influence ocular healtjh
* active ocular disease and no history of ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
difference in corneal sensitivity threshold baseline and after 7 days of extended contact lens wear | 7+/-1 days
  The difference in corneal sensitivity threshold baseline versus after 7 days of extended contact lens wear will be determined. Corneal sensitivity measurement will take place with the Swiss Liquid Jet Aesthesiometer for Corneal Sensitivity (SLACS) and will be recorded in mbar.

SECONDARY OUTCOMES:
correlation between corneal sensitvity threshold and subjective symptoms | 7+/-1 days
  correlation between corneal sensitvity threshold and subjective symptoms after 7 days of extended contact lens wear: corneal sensitivity threshold will be determinded with the Swiss Liquid Jet Aesthesiometer for Corneal Sensitivity (SLACS) and will be recorded in mbar. Subjective Symptoms will be recorded with the CLEDQ8 questionnaire (specifically designed to assess contact lens comfort)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Nosch, PhD, Principal Investigator — Institute of Optometry, FHNW
Locations (1):
- Institute of Optometry, Olten, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belmonte C, Acosta MC, Gallar J. Neural basis of sensation in intact and injured corneas. Exp Eye Res. 2004 Mar;78(3):513-25. doi: 10.1016/j.exer.2003.09.023. PMID 15106930
- [Background] Cheng KH, Leung SL, Hoekman HW, Beekhuis WH, Mulder PG, Geerards AJ, Kijlstra A. Incidence of contact-lens-associated microbial keratitis and its related morbidity. Lancet. 1999 Jul 17;354(9174):181-5. doi: 10.1016/S0140-6736(98)09385-4. PMID 10421298
- [Background] Morgan PB, Murphy PJ, Gifford KL, Gifford P, Golebiowski B, Johnson L, Makrynioti D, Moezzi AM, Moody K, Navascues-Cornago M, Schweizer H, Swiderska K, Young G, Willcox M. CLEAR - Effect of contact lens materials and designs on the anatomy and physiology of the eye. Cont Lens Anterior Eye. 2021 Apr;44(2):192-219. doi: 10.1016/j.clae.2021.02.006. Epub 2021 Mar 25. PMID 33775377
- [Background] Muller LJ, Marfurt CF, Kruse F, Tervo TM. Corneal nerves: structure, contents and function. Exp Eye Res. 2003 May;76(5):521-42. doi: 10.1016/s0014-4835(03)00050-2. PMID 12697417
- [Background] Nosch DS, Oscity M, Steigmeier P, Kaser E, Loepfe M, Joos RE. Working principle and relevant physical properties of the Swiss Liquid Jet Aesthesiometer for Corneal Sensitivity (SLACS) evaluation. Ophthalmic Physiol Opt. 2022 May;42(3):609-618. doi: 10.1111/opo.12962. Epub 2022 Feb 14. PMID 35156726